CLINICAL TRIAL: NCT06201754
Title: Association Between Bedside Air Quality in ICU and Complications Including Hospital Acquired Infections and Arrhythmia
Brief Title: Bedside Air Quality in ICU and Clinical Outcome
Status: Withdrawn | Type: Observational
Why Stopped: No Participants Enrolled
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Lingtong Huang, MD, Doctor, First Affiliated Hospital of Zhejiang University
Other Study IDs: IIT20230456B
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICU patients: We will include all ICU inpatients who undergo bedside air quality monitoring
  Interventions: Other: Measure air quality

INTERVENTIONS:
Other: Measure air quality — Measure air quality, including PM2.5、PM10

SUMMARY:
There is a close relationship between air pollution and cardiovascular disease. Small particulate matter and inhalable particulate matter in the air are the main components of air pollution, which can enter the respiratory system and enter the bloodstream through alveoli. These particles are believed to have the ability to trigger inflammatory responses, which are one of the important factors leading to cardiovascular disease. Some studies suggest that air pollution may increase the risk of cardiac events, such as arrhythmia and myocardial infarction, by affecting the autonomic function of the heart. Air pollution in the ICU may have a series of adverse effects on critically ill patients, especially those with underlying heart disease or elderly patients, but there is no relevant research to confirm this.

DETAILED DESCRIPTION:
Hospital acquired infections, also known as hospital acquired infections or healthcare related infections, refer to infections caused by activities related to treatment, diagnosis, or rehabilitation in the process of receiving medical services. Hospital acquired infections (HAIs) are a major global issue, and treatment may be costly. In the UK, it is estimated that as of 2017, the cost of HAIs could reach £ 1 billion per year, and hospital environments are considered to account for approximately 20% of all HAIs in terms of affecting the survival and transmission of pathogens in the environment. The hospital environment is influenced by workplace design and layout, operation and maintenance, as well as various interactions between the environment and people. Research on environmental microbial pollution indicates that various factors, including indoor air quality parameters (such as temperature, relative humidity, and ventilation), staff activities, patient conditions and visitor numbers, as well as surface types, may affect the presence of microorganisms. A very small amount of research associates virus concentration with these factors. The surfaces, air, and indoor structures including ventilation systems have been proven to serve as reservoirs for pathogens, and in some cases, these pathogens can survive for several months in hospital environments. Previous studies have utilized environmental sampling information to correlate air biomass levels, surface biomass, and HAIs incidence. Sampling of microorganisms in the air can be used to evaluate the concentration of microorganisms present in the hospital environment. Most studies use culture based methods to evaluate active microorganisms, and the microbial load in the air can be quantified using active or passive sampling methods.

The indoor air quality (IAQ) parameters in hospitals, including temperature, relative humidity, CO2 level (reflecting ventilation rate), particulate matter concentration, and particle size, are crucial for ensuring personnel health and may also affect the biological load in the environment. In indoor environments, temperature and relative humidity are the most commonly monitored indicators. However, these two parameters are associated with the survival of microorganisms, with humidity being a particularly noteworthy factor as many bacteria and fungi prefer humid environments. There is evidence to suggest that the survival rate of the virus increases when the relative humidity is below 40% RH. Although there are differences in guidance around the world, it is generally recommended to maintain room temperature between 16-25 ° C and humidity within the range of 40-60% RH. CO2 is related to the exhaled breath of relevant personnel and is often measured as an indicator of ventilation levels. Many studies have also shown that ventilation rates reflected by CO2 concentration can be used to assess the risk of airborne infections. The particulate matter in the air provides a general measure of indoor air quality (IAQ), which is related to indoor sources, activities, or outdoor conditions. Some studies suggest using particulate matter in the air as a monitoring indicator to measure air cleanliness, even when using ventilation systems in professional hospitals. The comprehensive consideration of these IAQ parameters can provide a more comprehensive understanding of the internal environmental conditions of the hospital, thereby helping to maintain the health and safety of patients and staff.

There is a close relationship between air pollution and cardiovascular disease. For a long time, scientific research has confirmed the adverse effects of air pollution on cardiovascular health. Small particulate matter (PM2.5) and inhalable particulate matter (PM10) in the air are the main components of air pollution, which can enter the respiratory system and enter the bloodstream through alveoli. These particles are believed to have the ability to trigger inflammatory responses, which are one of the important factors leading to cardiovascular disease. Some studies suggest that air pollution may increase the risk of cardiac events, such as arrhythmia and myocardial infarction, by affecting the autonomic function of the heart. Air pollution in the ICU may have a series of adverse effects on critically ill patients, especially those with underlying heart disease or elderly patients, but there is no relevant research to confirm this.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years old
2. The subject or their family members fully understand the patient's instructions and sign an informed consent form

Exclusion Criteria:

1. Expected ICU hospitalization days are less than 2 days
2. Pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study includes all patients in need of intensive care
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
PM2.5 exposures and hospital acquired infections | six month
  The correlation between the total amount or number of PM2.5 exposures (area under the curve and greater than 5ug/m3) and hospital acquired infections after admission to the ICU

SECONDARY OUTCOMES:
Air quality indicators and arrhythmias | six month
  Correlation between air quality indicators (PM2.5, PM10) and newly diagnosed arrhythmias
Medical operations and air quality indicators | six month
  Correlation between medical operations and air quality indicators (PM2.5, PM10)
PM10, CO2 and hospital acquired infections | six month
  Correlation between PM10 and hospital acquired infections
Air quality indicators and mechanical ventilation | six month
  Correlation between air quality indicators (PM2.5, PM10) and mechanical ventilation
Air quality indicators and the use of vasoactive drugs | six month
  Correlation between air quality indicators (PM2.5, PM10) and the use of vasoactive drugs
Air quality indicators and ventilator-associated pneumonia | six month
  Correlation between air quality indicators (PM2.5, PM10) and incidence rate of ventilator-associated pneumonia
Air quality indicators and incidence rate of CRBSI | six month
  Correlation between air quality indicators (PM2.5, PM10) and incidence rate of CRBSI

CONTACTS AND LOCATIONS:
Overall Officials: Lingtong Huang, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (3):
- China (3):
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First People's Hospital of Pinghu, Pinghu
  - Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University, Taizhou

IPD SHARING:
Plan to Share IPD: No